CLINICAL TRIAL: NCT00579280
Title: A Randomized, Double-blind, Placebo-controlled Study of Quetiapine SR and Divalproex Sodium ER on Anxiety in Bipolar Disorder With at Least Moderately Severe Current Anxiety and Lifetime Panic or Generalized Anxiety Disorder.
Brief Title: Quetiapine SR and Divalproex Sodium ER in the Treatment of Anxiety in Bipolar Disorder With Panic Disorder and/or GAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AZ 1107
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2012-07

CONDITIONS: Bipolar Disorder; Panic Disorder; Generalized Anxiety Disorder
Keywords: Randomized; Double-Blind; Placebo-Controlled; Quetiapine; DivalproexSodiumER; Bipolar; Anxiety; Panic; GAD
MeSH Terms: conditions — Bipolar Disorder; Panic Disorder; Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Quetiapine SR (Active Comparator): Quetiapine SR (Quetiapine Sustained Release)
  Interventions: Drug: quetiapine SR
- Divalproex Sodium ER (Active Comparator): Divalproex Sodium ER (Divalproex Sodium Extended Release)
  Interventions: Drug: divalproex sodium ER
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: quetiapine SR — flexible dosing, 50 mg up to a maximum of 300 mg per day for 8 weeks
  Arms: Quetiapine SR
Drug: divalproex sodium ER — Flexible dosing, 500 mg up to a maximum of 3000 mg per day for 8 weeks
  Arms: Divalproex Sodium ER
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
The specific aim of this study is to evaluate the efficacy, tolerability, and safety of quetiapine SR monotherapy and divalproex sodium ER monotherapy in comparison to placebo in the treatment of ambulatory bipolar disorder with co-morbid lifetime panic disorder or generalized anxiety disorder and current at least moderately severe anxiety.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, parallel-group, 8-week trial of quetiapine SR monotherapy compared to divalproex sodium ER monotherapy in outpatient subjects with a lifetime bipolar I, II, or not otherwsise specified (NOS) disorder, a lifetime panic or generalized anxiety disorder, and current diagnosis at least moderately severe anxiety symptoms. Approximately 180 subjects will be randomized to obtain 90 subjects who complete the 8-week trial (30 completers per treatment group). This calculation is based on drop out rates in a similar patient population carried out by this group of collaborators. Subjects will be randomized to quetiapine SR or divalproex sodium ER or placebo in a 1:1:1 ratio. No concomitant psychotropic medication will be allowed throughout the study except for prn lorazepam during the first two weeks for the management of affective and anxiety symptoms, prn zolpidem and zaleplon for the management of insomnia and benztropine for the management of extrapyramidal side effects (EPS). Throughout the study, psychiatric scales will be used to assess psychiatric symptoms and the presence of treatment-emergent adverse events will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age and not older than 65
* Subjects must have lifetime bipolar I, II, or not otherwise specified (NOS) disorder as defined by DSM-IV TR (Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision) criteria
* Subjects must have lifetime panic disorder or generalized anxiety disorder (GAD) as defined by DSM-IV, criteria (except clause "does not occur exclusively during a mood disorder" of Criterion F for GAD)
* Subjects' bipolar symptoms must be no more than moderate in severity, defined as a CGI-BP< 4
* Subjects' anxiety symptoms must be at least moderate in severity, defined as a CGI-S > 4
* Subjects must not be receiving regular mood stabilizing, antidepressant, antipsychotic, or anxiolytic medication for at least one week prior to baseline. Patients receiving fluoxetine or depot antipsychotics should be off these medications for at least four weeks prior to baseline
* Subjects or their legally authorized representative must sign the Informed Consent Document after the nature of the trial has been fully explained
* If female, subjects must be: postmenopausal, surgically incapable of childbearing, or practicing medically acceptable effective method(s) of contraception (e.g., hormonal methods, barrier methods, intrauterine device) for at least one month prior to study entry and throughout the study

Exclusion Criteria:

* Subjects who do not have lifetime bipolar disorder by DSM-IV-TR criteria
* Subjects who do not have lifetime panic disorder or generalized anxiety disorder by DSM-IV-TR criteria
* Subjects who are receiving treatment with an anti-manic or mood stabilizing medication (lithium, valproate, carbamazepine, or an antipsychotic), and in the investigators' judgment, require ongoing treatment with that medication
* Subjects whose bipolar symptoms are presently more than moderately severe (CGI-BP>5)
* Subjects whose anxiety symptoms are presently less than moderately severe (CGI-S<3)
* Subjects with clinically significant suicidal or homicidal ideation.
* Subjects with a current DSM-IV TR Axis I diagnosis of delirium, dementia, amnesia, or other cognitive disorders; a DSM-IV TR diagnosis of a substance dependence disorder within the past six months; a lifetime DSM-IV TR psychotic disorder (e.g., schizophrenia or schizoaffective disorder)
* Subjects with serious general medical illnesses including hepatic, renal, respiratory, cardiovascular, endocrine, neurological, or hematological disease as determined by the clinical judgment of the clinical investigator. Subjects with hypo-or hyperthyroidism unless stabilized on thyroid replacement > 3 months
* Subjects with a clinically significant abnormality in their pre-study physical exam, vital signs, EKG, or laboratory tests
* Subjects who are allergic to or who have demonstrated hypersensitivity or intolerance to either of the active study medications
* Women who are pregnant or nursing
* Subjects who have received an experimental drug or used an experimental device within 30 days
* Subjects who have a history of neuroleptic malignant syndrome
* A patient with diabetes mellitus (DM) fulfilling one of the following criteria:
* Unstable DM defined as enrollment glycosylated hemoglobin (HbAlc) >8.5%
* Admitted to hospital for treatment of DM or DM related illness within the past 12 weeks
* Not under physician care for DM
* Physician responsible for patient's DM care has not indicated that the patient's DM is controlled
* Physician responsible for patient's DM care has not approved the patient's participation in the study
* Has not been on the same dose of oral hypoglycemic drug(s) and/or diet for the 4 weeks before randomization. For thiazolidinediones (glitazones) this period should not be less than 8 weeks before randomization
* Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks Note: If a patient with DM meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Sheehan, MD, Principal Investigator — University of South Florida
Locations (3):
- United States (3):
  - VA Palo Alto HCS & Stanford School of Medicine, Palo Alto, California
  - University of South Florida College of Medicine, Tampa, Florida
  - University of Cincinnati Medical Center, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Quetiapine SR: Quetiapine SR (sustained release)
- Divalproex Sodium ER: Divalproex Sodium ER (extended release)
- Placebo: Placebo control
Period: Overall Study
Arm/Group | Quetiapine SR | Divalproex Sodium ER | Placebo
Started | 49 | 49 | 51
Completed | 47 (LOCF evaluable sample) | 46 (LOCF evaluable sample) | 51 (LOCF evaluable sample)
Not Completed | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine SR | Divalproex Sodium ER | Placebo | Total
Number analyzed (Participants) | 49 | 49 | 51 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 49 | 51 | 149
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.1) | 37.5 (12.0) | 37.6 (11.6) | 38.8 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 33 | 88
  Male | 21 | 22 | 18 | 61
Region of Enrollment [Number; unit: participants]
  United States | 49 | 49 | 51 | 149
Clinical Global Impression - Severity scale (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — Among the most wide used brief assessments in psychiatry, the Clinical Global Impression - Severity scale (CGI-S) is a measure of symptom severity for patients with psychiatric disorders. The range of response is from 1 (normal) through 7 (among the most severely ill patients). A higher score indicates greater severity.
  Reference Clinical Global Impression (CGI) Reference: Guy W, editor. Early Clinical Drug Evaluation (ECDEU) Assessment Manual for Psychopharmacology. 1976. Rockville, MD, U.S. Department of Health, Education, and Welfare
  units on a scale | 5.4 (.5) | 5.3 (.6) | 5.4 (.6) | 5.4 (.6)
Hamilton Anxiety Scale (HAM-A) [Mean (Standard Deviation); unit: units on a scale] — Hamilton Anxiety Scale (HAM-A) measures severity of anxiety symptoms. The range of scores is 0-56. Higher scores indicate worse anxiety.
  units on a scale | 41.4 (12.1) | 37.5 (12.0) | 37.6 (11.6) | 38.8 (12.0)
Sheehan Panic Disorder Scale (SPS) [Mean (Standard Deviation); unit: units on a scale] — Sheehan Panic Disorder Scale (SPS). The range of scores 0-140. A higher score indicates more severe symptoms of panic disorder.
  units on a scale | 47.5 (17.8) | 42.4 (18.5) | 41.8 (19.5) | 43.9 (18.7)
Montgomery Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — Montgomery Asberg Depression Rating Scale (MADRS) measures severity of depressive symptoms. The range of scores is 0-60. A higher score indicates worse depression.
  units on a scale | 26.4 (8.3) | 24.5 (7.3) | 25.8 (7.9) | 25.6 (7.8)
Young Mania Rating Scale (YMRS) [Mean (Standard Deviation); unit: units on a scale] — Young Mania Rating Scale (YMRS) measures severity of mania / hypomania symptoms. The range of scores is 0-60. A higher score indicates worse mania / hypomania.
  units on a scale | 11.2 (6.1) | 12.3 (7.9) | 11.2 (5.7) | 11.6 (6.6)
Sheehan Disability Scale (SDS) [Mean (Standard Deviation); unit: units on a scale] — Sheehan Disability Scale (SDS) measures severity of functional impairment or disability. There are 4 scores: 1) Work Disability 2) Social Disability 3) Family Life Disability. Each of these domains is scored 0-10, with a higher score representing greater disability or functional impairment. These 3 domain scores are added to give a Total Disability scale score. On total disability the score ranges from 0 to 30, with a higher score representing greater total disability or functional impairment.
  units on a scale | 15.1 (6.8) | 12.9 (7.9) | 14.8 (7.4) | 14.3 (7.4)
Rapid Ideas Scale [Mean (Standard Deviation); unit: units on a scale] — Rapid ideas Scale (RISc) measures severity of rapid thoughts - range of scores 0-100 - the higher score represents more severe rapidity of thinking.
  units on a scale | 54.0 (17.3) | 52.1 (20.9) | 51.7 (19.1) | 52.6 (19.1)
Sheehan Irritability Scale (SIS) [Mean (Standard Deviation); unit: units on a scale] — Sheehan Irritability Scale (SIS) measures severity of anxiety symptoms. The range of scores is 0-70. A higher score indicates worse irritability.
  units on a scale | 48.9 (11.5) | 43.2 (16.4) | 43.5 (13.9) | 45.2 (14.2)
Suicidality Tracking Scale [Mean (Standard Deviation); unit: units on a scale] — Sheehan - Suicidality Tracking Scale (S-STS) (2008 version with 8 items) measures severity of a range of suicidality symptoms. Range of scores: 0-32. A higher score represents more severe suicidality. Population: This scale was only administered to the last 74 patients in the trial
  units on a scale
    number analyzed (Participants) | 19 | 28 | 27 | 74
    (all) | 1.9 (2.6) | 1.8 (2.8) | 1.0 (1.5) | 1.5 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the CGI-21 Anxiety
Description: The CGI-21 Anxiety is a 21-point clinician-rated global improvement for anxiety symptoms. Response range: -10 to +10. The higher the score the more improvement. At Baseline all patients have a score of "0" (zero), against which any subsequent improvements or deterioration is assessed. The relative efficacy of the 3 treatments was tested with a last-observation-carried forward (LOCF) repeated-measures analysis of variance (ANOVA). The focus was on the "treatment-by-time" effect showing whether the trajectory of response differed over time by treatment group. Also, group differences in baseline-to-endpoint changes in the efficacy measure were tested using LOCF ANOVA followed by pairwise planned comparisons (t-tests). The least square means shown here are from the LOCF baseline-to-endpoint ANOVA. Outcomes showing scores above zero indicate that patients did better, i.e. showed improvement on this scale.
Time Frame: 8 weeks (using LOCF Repeated Measures ANOVA)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Quetiapine SR: Quetiapine SR
  quetiapine SR: flexible dosing, 50 mg up to a maximum of 300 mg per day for 8 weeks
- Divalproex Sodium ER: Divalproex Sodium ER
  divalproex sodium ER: Flexible dosing, 500 mg up to a maximum of 3000 mg per day for 8 weeks
Arm/Group | Quetiapine SR | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 47 | 46 | 51
score on a scale | 4.9 (0.62) | 2.9 (0.63) | 3.4 (0.60)
Statistical Analysis 1: Comparison: Quetiapine SR vs Divalproex Sodium ER vs Placebo; Test type: Superiority; p < .05, ANOVA

2. Secondary Outcome: Change From Baseline on Patient Global Improvement Scale (PGI-21) for Anxiety Symptoms
Description: The PGI-21 Anxiety is a 21-point patient-rated global improvement for anxiety symptoms. Response range: -10 to +10. The higher the score the more improvement. At Baseline all patients have a score of "0" (zero), against which any subsequent improvements or deterioration is assessed. The relative efficacy of the 3 treatments was tested with a last-observation-carried forward (LOCF) repeated-measures analysis of variance (ANOVA). The focus was on the "treatment-by-time" effect showing whether the trajectory of response differed over time by treatment group. Also, group differences in baseline-to-endpoint changes in the efficacy measure were tested using LOCF ANOVA followed by pairwise planned comparisons (t-tests). The least square means shown here are from the LOCF baseline-to-endpoint ANOVA. Outcomes showing scores above zero indicate that patients did better, i.e. showed improvement on this scale.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine SR | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 47 | 46 | 51
score on a scale | 3.9 (0.68) | 1.9 (0.69) | 2.3 (0.65)
Statistical Analysis 1: Comparison: Quetiapine SR vs Divalproex Sodium ER vs Placebo; Test type: Superiority; p < 0.05, ANOVA

3. Secondary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) Scores
Description: Hamilton Anxiety Scale (HAM-A) measures severity of anxiety symptoms - range of scores is 0-56. A higher score means worse anxiety. The relative efficacy of the 3 treatments was tested with a last-observation-carried forward (LOCF) repeated-measures analysis of variance (ANOVA) in which baseline and each of the 8 weekly assessments were the within subject factors (labeled "time") and treatment group (labeled "treatment") was the between-subjects factor with 3 levels. The focus was on the "treatment-by-time" effect showing whether the trajectory of response differed over time by treatment group. Also, group differences in baseline-to-endpoint changes in the efficacy measure were tested using LOCF ANCOVA followed by pairwise planned comparisons (t-tests). The least square means shown here are from the LOCF baseline-to-endpoint ANCOVA. Outcome results with a "minus" score indicate that patients did better, i.e. had a reduction in symptoms on this scale.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine SR | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 47 | 46 | 51
score on a scale | -11.7 (1.32) | -6.4 (1.30) | -8.4 (1.4)
Statistical Analysis 1: Comparison: Quetiapine SR vs Divalproex Sodium ER vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

4. Secondary Outcome: Change From Baseline in Sheehan Panic Disorder Scale (SPS)
Description: Sheehan Panic Disorder Scale (SPS). Range of scores: 0-140. Higher scores indicate greater severity of symptoms. The relative efficacy of quetiapine SR vs. divalproex ER and placebo was tested using a last-observation-carried forward (LOCF) repeated-measures analysis of variance (ANOVA) in which baseline and each of the 8 weekly assessments for the efficacy variables were the within subject factors ("time") and treatment group ("treatment") was the between-subjects factor with 3 levels. The focus in this analysis was on the "treatment-by-time" effect showing whether the trajectory of response differed over time by treatment group. Also, group differences in baseline-to-endpoint changes in efficacy measures were tested using LOCF ANCOVA followed by pairwise planned comparisons (t-tests). The least square means shown here are from the baseline-to-endpoint LOCF ANCOVA. Outcome results with a "minus" indicate that patients did better, i.e. had a reduction in symptoms on this scale.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine SR | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 47 | 46 | 51
score on a scale | -24.4 (2.9) | -14.8 (2.9) | -18.3 (2.8)
Statistical Analysis 1: Comparison: Quetiapine SR vs Divalproex Sodium ER vs Placebo; Test type: Superiority; p < .05, ANCOVA

5. Secondary Outcome: Change From Baseline on Montgomery Asberg Depression Rating Scale (MADRS)
Description: Montgomery Asberg Depression Rating Scale (MADRS) measures severity of depressive symptoms. Range of scores: 0-60. A higher score shows greater severity of depressive symptoms. The relative efficacy of the 3 treatments was tested with a last-observation-carried forward (LOCF) repeated-measures analysis of variance (ANOVA) in which baseline and each of the 8 weekly assessments were the within subject factors ("time") and treatment group ("treatment") was the between-subjects factor with 3 levels. The central focus was on the "treatment-by-time" effect showing whether the trajectory of response differed over time by treatment group. Also, group differences in baseline-to-endpoint changes in efficacy were tested using LOCF ANCOVA followed by pairwise planned comparisons (t-tests). The least square means shown here are from the LOCF baseline-to-endpoint ANCOVA. Outcome results with a "minus" score indicate that patients did better, i.e had a reduction in symptoms on this scale.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine SR | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 47 | 46 | 51
score on a scale | -11.5 (1.5) | -5.5 (1.6) | -7.3 (1.5)
Statistical Analysis 1: Comparison: Quetiapine SR vs Divalproex Sodium ER vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

6. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS)
Description: Young Mania Rating Scale (YMRS) measures severity of mania / hypomania symptoms. Range of scores: 0-60. A higher score shows worse mania / hypomania. The relative efficacy of the 3 treatments was tested with a last-observation-carried forward (LOCF) repeated-measures analysis of variance (ANOVA) in which baseline and each of the 8 weekly assessments were the within subject factors ("time") and treatment group ("treatment") was the between-subjects factor with 3 levels. The focus was on the "treatment-by-time" effect showing whether the trajectory of response differed over time by treatment group. Also, group differences in baseline-to-endpoint changes in the efficacy measure were tested using LOCF ANCOVA followed by pairwise planned comparisons (t-tests). The least square means shown here are from the LOCF baseline-to-endpoint ANCOVA. Outcome results with a "minus" score indicate that patients did better, i.e. had a reduction in symptoms on this scale.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine SR | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 47 | 46 | 51
score on a scale | -5.4 (1.2) | -4.4 (1.2) | -4.3 (1.1)
Statistical Analysis 1: Comparison: Quetiapine SR vs Divalproex Sodium ER vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

7. Secondary Outcome: Change From Baseline on Clinician Global Impression Scale for Bipolar Disorder (CGI-BP) (Overall Severity)
Description: Clinician Global Impression Scale for Bipolar Disorder (CGI-BP) measures the severity of bipolar disorder symptoms overall. Range of response: i1. normal, not ill to 7. very severely ill. A higher score represents greater severity. A last-observation-carried forward (LOCF) repeated-measures analysis of variance (ANOVA) in which baseline and each of the 8 weekly assessments were the within subject factors ("time") and treatment group ("treatment") was the between-subjects factor with 3 levels was used. The focus was on the "treatment-by-time" effect and whether the trajectory of response differed over time by treatment. Also, group differences in baseline-to-endpoint changes in the efficacy measure were tested using LOCF ANCOVA followed by pairwise planned comparisons (t-tests). The least square means shown here are from the LOCF baseline-to-endpoint ANCOVA. Outcome results with a "minus" score indicate that patients did better, i.e. had a reduction in symptoms on this scale.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine SR | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 47 | 46 | 51
score on a scale | -1.2 (.16) | -.5 (.17) | -1.0 (.16)
Statistical Analysis 1: Comparison: Quetiapine SR vs Divalproex Sodium ER vs Placebo; Test type: Superiority; p < 0.05, Chi-squared; Differences in response (70% or greater improvement) and remission (50% or greater improvement) rates between the groups

8. Secondary Outcome: Change From Baseline on Rapid Ideas Scale (RISc)
Description: Rapid ideas Scale (RISc) measures severity of rapid thoughts. Range of scores is 0-100. A higher score means more severe rapidity of thinking. The relative efficacy of the 3 treatments was tested with a last-observation-carried forward (LOCF) repeated-measures analysis of variance (ANOVA) in which baseline and each of the 8 weekly assessments were the within subject factors ("time") and treatment group ("treatment") was the between-subjects factor with 3 levels. The focus was on the "treatment-by-time" effect showing whether the trajectory of response differed over time by treatment group. Also, group differences in baseline-to-endpoint changes in the efficacy measure were tested using LOCF ANCOVA followed by pairwise planned comparisons (t-tests). The least square means shown here are from the LOCF baseline-to-endpoint ANCOVA. Outcome results with a "minus" score indicate that patients did better, i.e. had a reduction in symptoms on this scale.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine SR | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 47 | 46 | 51
score on a scale | -28.9 (3.4) | -19.7 (3.4) | -23.1 (3.3)
Statistical Analysis 1: Comparison: Quetiapine SR vs Divalproex Sodium ER vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

9. Secondary Outcome: Change From Baseline in Sheehan Irritability Scale (SIS)
Description: Sheehan Irritability Scale (SIS) measures severity of anxiety symptoms. Range of scores: 0-70. A higher score shows worse irritability. The relative efficacy of the 3 treatments was tested with a last-observation-carried forward (LOCF) repeated-measures analysis of variance (ANOVA) in which baseline and each of the 8 weekly assessments were the within subject factors ("time") and treatment group ("treatment") was the between-subjects factor with 3 levels. The focus was on the "treatment-by-time" effect showing whether the trajectory of response differed over time by treatment group. Also, group differences in baseline-to-endpoint changes in the efficacy measure were tested using LOCF ANCOVA followed by pairwise planned comparisons (t-tests). The least square means shown here are from the LOCF baseline-to-endpoint ANCOVA. Outcome results with a "minus" score indicate that patients did better, i.e. had a reduction in symptoms on this scale.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine SR | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 47 | 46 | 51
score on a scale | -29.8 (3.4) | -22.6 (3.4) | -19.4 (3.3)
Statistical Analysis 1: Comparison: Quetiapine SR vs Divalproex Sodium ER vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

10. Secondary Outcome: Change From Baseline on Sheehan Disability Scale (SDS) - Total
Description: Sheehan Disability Scale (SDS) measures severity of functional impairment or disability. There are 4 scores: 1) Work Disability 2) Social Disability 3) Family Life Disability. Each of these domains is scored 0-10, with a higher score representing greater disability or functional impairment. These 3 domain scores are added to give a Total Disability scale score. Range of response for Total Disability: 0 to 30. A higher score shows greater disability/functional impairment. The relative efficacy of the 3 treatments was tested with a last-observation-carried forward (LOCF) repeated-measures analysis of variance (ANOVA). Also, group differences in baseline-to-endpoint changes in the efficacy measure were tested using LOCF ANCOVA followed by pairwise planned comparisons (t-tests). The least square means shown here are from the LOCF baseline-to-endpoint ANCOVA. Outcome results with a "minus" score indicate that patients did better, i.e. had a reduction in symptoms on this scale.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine SR | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 47 | 46 | 51
score on a scale | -6.5 (1.8) | -3 (1.2) | -5.3 (1.1)
Statistical Analysis 1: Comparison: Quetiapine SR vs Divalproex Sodium ER vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

11. Secondary Outcome: Change From Baseline on Sheehan- Suicidality Tracking Scale S-STS (2008 Version With 8 Items)
Description: Sheehan - Suicidality Tracking Scale S-STS (2008 version with 8 items) measures severity of a range of suicidality symptoms. Range of scores: 0-32. A higher score represents more severe suicidality. The relative efficacy of the 3 treatments was tested with a last-observation-carried forward (LOCF) repeated-measures analysis of variance (ANOVA) in which baseline and each of the 8 weekly assessments were the within subject factors ("time") and treatment group ("treatment") was the between-subjects factor with 3 levels. Also, group differences in baseline-to-endpoint changes in the efficacy measure were tested using LOCF ANCOVA followed by pairwise planned comparisons (t-tests). The least square means shown here are from the LOCF baseline-to-endpoint ANCOVA. Outcome results with a "minus" score indicate that patients did better, i.e. had a reduction in symptoms on this scale..
Time Frame: 8 weeks
Population: Only administered to the last 74 patients enrolled after November 2008
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Quetiapine SR | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 19 | 28 | 27
score on a scale | -.95 (.44) | -.07 (.36) | -.3 (.38)
Statistical Analysis 1: Comparison: Quetiapine SR vs Divalproex Sodium ER vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

ADVERSE EVENTS:
Arm/Group | Quetiapine SR | Divalproex Sodium ER | Placebo
Serious Adverse Events (participants affected / at risk) | 1/49 | 3/49 | 2/51
Other Adverse Events (participants affected / at risk) | 24/49 | 18/49 | 17/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine SR (N=49) | Divalproex Sodium ER (N=49) | Placebo (N=51)
fainted (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
spider bite (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
worsening depression (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine SR (N=49) | Divalproex Sodium ER (N=49) | Placebo (N=51)
Drowsiness/Sleepiness (Nervous system disorders) | 24 | 18 | 17
Dry Mouth (Gastrointestinal disorders) | 15 | 3 | 7
Nausea or Nausea/Vomiting (Gastrointestinal disorders) | 9 | 12 | 14
Tingling (Skin and subcutaneous tissue disorders) | 8 | 1 | 1
Increased appetite (Gastrointestinal disorders) | 7 | 6 | 7
Sedation (Nervous system disorders) | 6 | 3 | 3
Headache (Nervous system disorders) | 4 | 12 | 12
Lightheadednessa (Nervous system disorders) | 4 | 2 | 1
Tiredness (Nervous system disorders) | 3 | 1 | 3
Diarrheaa (Gastrointestinal disorders) | 1 | 2 | 4
Dizzinessa (Nervous system disorders) | 1 | 3 | 1

LIMITATIONS AND CAVEATS:
Study was limited to 8 weeks and to patients with bipolar disorder and comorbid panic disorder or generalized anxiety disorder.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes